CLINICAL TRIAL: NCT04464369
Title: Functional Dyspepsia: Validation of a Questionnaire for Symptom Assessment in Patients Suffering From Post Prandial Distress Syndrome (Functional Dyspepsia) :
Brief Title: Functional Dyspepsia: Validation of the Leuven Postprandial Distress Scale (LPDS) in a Placebo-controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: S54963
Record Dates: First submitted 2016-04-08; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Functional Dyspepsia
Keywords: functional dyspepsia; postprandial distress syndrome
MeSH Terms: interventions — itopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo t.i.d.
  Interventions: Drug: Placebo
- Itopride (Active Comparator): Itopride co 100 mg t.i.d.
  Interventions: Drug: itopride

INTERVENTIONS:
Drug: itopride — itopride is a gastroprokinetic drug that has previously been evaluated in the treatment of functional dyspepsia and which is available in a number of countries worldwide
  Other Names: Ganaton
  Arms: Itopride
Drug: Placebo — placebo pills matching the look and weight of the itopride tablets
  Arms: Placebo

SUMMARY:
No instrument is available for the assessment of the symptoms in patients suffering from functional dyspepsia - postprandial distress syndrome patients - PDS. Indeed PDS is an unmet clinical need in drug development. To do so, the development of suitable endpoints for its efficacy evaluation is indicated.

After interviews of patients suffering from PDS (Focus groups) and identification of the emerging symptoms a draft version of the Leuven Postprandial Distress Scale (LPDS) questionnaire has been designed. This study will assess the reliability of the scoring rule, the construct validity and ability to detect change of the draft LPDS.

A minimum of 100 PDS patients will be randomised in two arms receiving respectively either Itopride 100 mg tid or Placebo tid during 8 weeks. Patients of both arms will be tested with LPDS using daily diary cards and by anchor questionnaires (PAGI-SYM, OSS, OTE) at baseline and during the study drug administration period.

DETAILED DESCRIPTION:
2.3 Study design After review of the literature, identification of the intended population (PDS patients with the lowest EPS component), it has been decided that the conceptual framework for the instrument will be based on the motility subscales of DSSI assessing the severity of the symptoms on 5 point Likert Scale (0-4; no symptom, mild, moderate, severe, very severe). After interview of patients suffering from PDS (Focus groups) and identification of the emerging symptoms a draft version of LPDS questionnaire has been designed. This study will assess the reliability of the scoring rule, the construct validity and ability to detect change of the draft LPDS.

A minimum of 100 PDS patients will be randomised in two arms receiving respectively either Itopride 100 mg tid or Placebo tid during 8 weeks. Patients of both arms will be tested with LPDS using daily diary cards and by PAGI-SYM, SF-NDI, OSS, OTE at baseline and during the study drug administration period.

Eligibility (2w) Randomisation Study drug administration (8w)

Group 1 Placebo tid (LPDS, OTE, OSS, PAGI-SYM, SF-NDI) Eligible patients Group 2 Itopride 100 mg tid (LPDS, OTE, OSS, PAGI-SYM, SF-NDI)

4.1 Interventional study for LPDS responsiveness. This study will be a multicentre randomized multiple-assessed, placebo-controlled parallel-group study of Itopride 100 mg tid in PDS. The rationale to use Itopride is the lack of efficient treatment for FD. Itopride was extensively used in FD trials and is prescribed in clinical practice in several parts of the world. The treatment period for evaluation of LPDS responsiveness will be 8 weeks after a 2 week eligibility period.

Patients will assess the severity of their symptoms using the new LPDS questionnaire adapted from the conceptual framework. This will be done through daily paper diaries. Assumingly, the diaries will include ratings of PDS symptoms, EPS symptoms, bloating, nausea and belching. In addition, patients will fill out OSS, PAGI-SYM and SF-NDI questionnaires at the end of the run-in period, and after 2, 4, 6 and 8 weeks of treatment. They will also fill out OTE after 2, 4, 6 and 8 weeks of treatment. (See these different questionnaires and the rationale to use them in annex)

At the end of the study, patients will be proposed to enter an open label period of one month (Itopride 100 mg tid). This open label period is not part of the study and has been associated for the benefit of the patients.

4.2 Assessment of symptom severity

Individual symptom severity (hypothesized for LPDS) will be assessed in daily diaries using a 5-point Likert scale:

0 - No symptom

1. - Mild (Symptom is present but is not bothersome)
2. - Moderate (Symptom is present and bothersome)
3. - Severe (Symptom interferes with normal activity)
4. - Very severe (Normal activity is not possible)

Overall symptom severity assessment (OSS) questionnaire (with 1 week recall):

What was the overall severity of your stomach symptoms during the past week? (Please select one answer)

* No symptoms
* Very mild
* Mild
* Moderate
* Severe
* Very severe

Overall Treatment Evaluation (OTE) questionnaire (with 1 week recall):

When thinking about the last week, how have your stomach symptoms have been (compared to your condition before you started this treatment)? (please select one answer)

* Extremely better
* Much better
* Somewhat better
* A little better
* About the same
* A little worse
* Somewhat worse
* Much worse
* Extremely worse

PAGI-SYM and SF-NFI are more complex and described in the literature

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for randomisation if all of the following criteria are met:

At visit 1:

1. Patients with FD diagnosis as per Rome III classification (Negative gastroscopy valid for the last 6 months)
2. Patients with PDS diagnosis as per Rome III by Rome III questionnaire
3. Patients must provide witnessed written informed consent prior to any study procedures being performed
4. Patients who are HP negative provided that they where not eradicated during the last 3 months.
5. Patients aged between 18 and 70 years inclusive
6. Male or female patients
7. Patients who are capable to understand the study and the questionnaires, and to comply with the study requirements

   At visit 2:
8. Patients suffering from active PDS (Rome III) as per LPDS scoring system (See Focus Group study) during 2 weeks before randomisation

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria are met:

At visit 1:

1. Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for entry into the study
2. Patients with any major psychiatric disorder (including those with a major psychosomatic element to their gastrointestinal disease), depression, alcohol or substance abuse in the last 2 years. Patients suffering from one psychiatric trouble stabilised for six month by the administration of one drug (Not amitryptiline) are acceptable.
3. Females who are pregnant or lactating.
4. Patients presenting with predominant symptoms of irritable bowel syndrome (IBS)
5. Patient with predominant symptoms of GERD according to GERD questionnaire (Two "yes" answer to question 21)
6. Patients suffering from diabetes type 1 or type 2.
7. Patients taking medications for the treatment of their upper digestive symptoms: prokinetics and acid suppressants (PPIs). A wash-out is allowed if medically indicated (E.g.: lack of efficacy or side-effects). This wash-out is minimum two weeks for the patients taking PPIs*
8. Patients with well-known hypersensitivity to gastroprokinetic drugs.
9. Patients with confirmed gastro-intestinal disease.
10. Patients with former digestive surgery affecting the gut motility.

    * Many patients take PPIs in absence of efficient treatment. In the literature, PPIs appear effective in patients suffering from substantial concomitant heartburn that is not allowed for inclusion in this study. In this context, a medically indicated wash-out and the proposal of a therapeutic alternative is appropriate.

6. Patients presenting symptoms of EPS several times a week according to Rome III questionnaire (score 5 on question 10) at visit 2

7. Patients presenting daily symptoms of CIN on Rome III questionnaire (score 6 on question 6 or score 5 on question 9) at visit 2

8. Patients presenting daily symptoms of Excessive belching according to Rome III questionnaire (score 6 on question 19) at visit 2

At visit 2:

1. Patients presenting symptoms of EPS several times a week according to Rome III questionnaire (score 5 on question 10)
2. Patients presenting daily symptoms of CIN on Rome III questionnaire (score 6 on question 6 or score 5 on question 9 )
3. Patients presenting daily symptoms of Excessive belching according to Rome III questionnaire (score 6 on question 19)
4. Patients presenting predominant GERD according to GERD questionnaire (Two"yes" answer to question 21)
5. Patients taking prohibited medications.
6. Patients affected by concomitant disease responsible for digestive symptoms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Responsiveness of the LPDS instrument (LPDS vs. PAGI-SYM) | 8 weeks
  The responsiveness of the LPDS will be evaluated in several ways. The correlation between changes in LPDS scores and changes in the (fullness/early satiation subscales of the) PAGI-SYM.
Responsiveness of the LPDS instrument (LPDS vs. PAGI-Qol) | 8 weeks
  The responsiveness of the LPDS will be evaluated in several ways. The correlation between changes in LPDS scores and changes in the the PAGI-QOL.
Responsiveness of the LPDS instrument (LPDS vs. OTE) | 8 weeks
  Changes in the LPDS scores from baseline to week 2 and week 4 will be correlated with the OTE at week 2 and 4
Responsiveness of the LPDS instrument (known-groups validation) | 8 weeks
  groups of patients will be formed on the basis of changes in OSS ratings over time, and changes in LPDS scores will be compared across these groups and the significance of the difference in mean changes in LPDS will be tested using analysis of variance

SECONDARY OUTCOMES:
The reliability of the LPDS instrument | Week 8
  The reliability of the LPDS instrument will be evaluated using internal consistency methods, by computing Cronbach's alpha coefficient from the correlation among the symptom items using data from different time points throughout the study. In addition, the test-retest reliability will be evaluated by correlating scores between days 1 and 4 during the run-in period.
Validity of the LPDS instrument | Week 8
  The construct validity of the LPDS will be tested using the logic of known-groups validity. This approach compares the mean scores from LPDS across groups known to differ on the patient's assessment of OSS and OTE. The significance of the difference in mean LPDS will be tested using analysis-of-variance methods.

OTHER OUTCOMES:
Effiacy of itopride | Week 8
  After blinded analysis for validation of the LPDS instrument the code will be broken and efficacy of itopride versus placebo will be evaluated using the LPDS instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, M.D., Ph.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tack J, Talley NJ, Camilleri M, Holtmann G, Hu P, Malagelada JR, Stanghellini V. Functional gastroduodenal disorders. Gastroenterology. 2006 Apr;130(5):1466-79. doi: 10.1053/j.gastro.2005.11.059. PMID 16678560
- Available data/document: Study Protocol: LPDSItopride study — http://www.targid.eu